CLINICAL TRIAL: NCT01596751
Title: Enhancing Efficacy of Chemotherapy in Triple Negative/Basal-Like Breast Cancer by Targeting Macrophages: A Multicenter Phase Ib/II Study of PLX 3397 and Eribulin in Patients With Metastatic Breast Cancer
Brief Title: Phase Ib/II Study of PLX 3397 and Eribulin in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hope Rugo, MD (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); Plexxikon (Industry)
Responsible Party: Sponsor-Investigator, Hope Rugo, MD, Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 12751; NCI-2015-01321 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2012-05-07; First posted 2012-05-11 (Estimated); Results first posted 2020-05-14 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic; breast; cancer; triple; negative; PLX; Eribulin
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — pexidartinib; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase Ib: 600 mg/Day PLX3397 Combined with Eribulin (Experimental): Treatments are given in 21 day cycles. For each cycle, treatment includes:
  * PLX3397 at a dose of 600 mg/day taken by mouth in the form of 100-200 mg gelcaps
  * Eribulin at dose of 1.4 mg/m2 given intravenously on days 1 and 8.
  Interventions: Drug: PLX3397; Drug: Eribulin
- Phase Ib: 800 mg/Day PLX3397 Combined with Eribulin (Experimental): Treatments are given in 21 day cycles. For each cycle, treatment includes:
  * PLX3397 at a dose of 800 mg/day taken by mouth in the form of 100-200 mg gelcaps
  * Eribulin at dose of 1.4 mg/m2 given intravenously on days 1 and 8
  Interventions: Drug: PLX3397; Drug: Eribulin
- Phase Ib: 1000 mg/Day PLX3397 Combined with Eribulin (Experimental): Treatments are given in 21 day cycles. For each cycle, treatment includes:
  * PLX3397 at a dose of 1000 mg/day taken by mouth in the form of 100-200 mg gelcaps
  * Eribulin at dose of 1.4 mg/m2 given intravenously on days 1 and 8
  Interventions: Drug: PLX3397; Drug: Eribulin
- Phase II: 800 mg/Day PLX3397 Lead in +Combined with Eribulin (Experimental): Treatment begins with a 7 day Lead-in phase of PLX3397 alone, followed by 21 day cycles of PLX3397 in combination with eribulin.
  Lead-in phase treatment:
  * PLX3397 at a dose of 800 mg/day given by mouth in the form of 100-200 mg gelcaps for 5 days followed by 2 days of rest.
  Treatment given in each 21 day cycle:
  * PLX3397 at a dose of 800 mg/day given by mouth in the form of 100-200 mg gelcaps for 5 days followed by 2 days of rest, repeated weekly
  * Eribulin at dose of 1.4 mg/m2 given intravenously on days 1 and 8
  Interventions: Drug: PLX3397; Drug: Eribulin

INTERVENTIONS:
Drug: PLX3397 — Dosage Form: 100 mg or 200 mg capsules, Dosage: 400 - 1000 mg, oral administration
Drug: Eribulin — Dosage Form: 1 mg per 2 mL (0.5 mg per mL); Solution (clear, colorless, sterile, packaged in glass vial) Dosage: 1.4 mg/m2, 2-5 min IV, Day 1, 8 q21 days
  Other Names: Halaven; E7389

SUMMARY:
The purpose of the Phase 1b portion of the study is to determine the best dose of PLX3397 when given in combination with standard dose eribulin (Halaven™). The purpose of the Phase 2 portion of the study is to find out what effects, good and/or bad, these drugs have on patients and their metastatic breast cancer.

DETAILED DESCRIPTION:
This is a nonrandomized, open label phase Ib/II study evaluating the safety and efficacy of eribulin in combination with PLX3397, a novel CSF1 inhibitor, in patients with metastatic breast cancer. The phase II portion of this trial will be limited to patients with triple negative disease.

The phase I portion of this trial is a dose escalation of PLX3397 to determine the maximum tolerated dose (MTD) of PLX3397 when given in combination with standard dose eribulin. Patients will be enrolled in cohorts of three, using the dose levels and plan outlined in the statistical section, with 6 patients enrolled at the MTD. All patients with accessible tumor will be required to have a tumor biopsy at study start before starting therapy. Pharmacokinetics of PLX3397 and eribulin, and blood levels of CSF1 will be obtained as outlined in section 14. To allow rapid accrual to phase Ib, and an earlier start to the phase II trial, patients will be enrolled in phase I with both hormone receptor positive and negative disease, and at any line of therapy assuming eligibility criteria are otherwise met.

Dose limiting toxicity (DLT) will be defined as any treatment-related toxicity meeting the criteria below and occurring within the first 21 days of combination therapy. Patients must receive at least 14 days of PLX3397 and 2 doses of eribulin during the first cycle in order to be considered evaluable for DLT (unless the missed doses are due to a DLT).

Patients in each cohort will be followed for at least 3 weeks (one full cycle) before opening accrual to the next dose level. If one patient in any cohort develops a DLT, an additional 3 patients will be enrolled at that level. If no additional toxicities occur in the six patients, then this particular dose would be used for the phase II trial, and the next higher dose would be considered the MTD. A minimum of 12 and maximum of 24 patients will be enrolled in the phase I study. The phase II trial will not open until the last patient in the phase I study has been followed for at least 3 weeks.

The phase II portion of this trial will evaluate progression free survival (PFS) in patients with Triple negative breast cancer (TNBC) treated with PLX3397 and eribulin, using the dose of PLX3397 determined in the phase Ib study in a two-step design. Please see the statistical section for details regarding enrollment and statistical design. Treatment is preceded by a 5 to 7 day lead-in phase, in which patients will take PLX3397 alone daily. Patients with accessible tumor will undergo a core biopsy of tumor before the start of PLX3397 treatment, and then a fine needle aspiration or core biopsy will be performed on the day of or the day before the start of eribulin (day -1 to day 0).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of breast cancer with documented progressive disease.
* Patients with stable brain metastases are eligible for this trial.
* At least one prior chemotherapy regimen for metastatic breast cancer. Prior treatment must be discontinued at least 2 weeks before treatment start.
* Concomitant therapy with bisphosphonates is allowed.
* Stable dose coumadin anticoagulation is allowed, providing that anticoagulation can be safely held to an International Normalized Ratio (INR) within normal range for the purpose of tumor biopsy. Low molecular weight heparin (LMWH is the preferred method of anticoagulation.
* Prothrombin time (PT)/International Normalized Ratio (INR) and partial thromboplastin time (PTT) within institutional normal limits within two weeks before initial biopsy.
* Measurable disease, as defined by RECIST guidelines or evaluable disease. Bone metastases must be evaluable.
* Disease amenable to core biopsy. Patients with pulmonary metastases as their only site of disease may enroll on this trial and will not undergo biopsy.
* For Phase I: patients with human epidermal growth factor receptor 2 (HER2) overexpressing disease must have been previously treated with trastuzumab. Patients with HER2 overexpressing disease are not eligible for the Phase II trial.
* Age eighteen years or older.
* Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
* Life expectancy of >/= 12 weeks.
* Patients with < grade 1 peripheral neuropathy are eligible for this trial.
* Adequate bone marrow reserve: Absolute Neutrophil Count (ANC) >/= 1000, platelets >/= 100,000.
* Adequate renal function: serum creatinine </= 1.5x upper limit of normal (ULN) OR calculated creatinine clearance ≥ 50 ml/min.
* Sodium, potassium, and chloride levels within institutional normal limits.
* Adequate hepatic function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) </= 2.5 x ULN, and total bilirubin </= 1.5x upper limit of normal. In patients with liver dysfunction due to hepatic metastases, AST and ALT are permitted to be </= 5 times the ULN.
* At baseline: Ejection fraction (EF) ≥ 50%, no evidence of QT prolongation, no history of congenital long QT syndrome, and no use of drugs known to increase the risk of Torsades de Point - patients may be eligible for study if the drug can be changed to another agent with less risk (such as changing from citalopram to an alternate antidepressant).
* Able to take oral medications and maintain hydration.
* Ability to give written informed consent and willingness to comply with the requirements of the protocol
* Women of child-bearing potential must agree to use an effective method of birth control during treatment and for six months after receiving their last dose of study drug

Specific inclusion criteria for Phase II

• Patients enrolling on the phase II portion of this trial must have ER, progesterone receptors (PR) and HER2 negative disease defined as less than 10% staining for ER and PR, and HER2 not amplified byFluorescent in situ hybridization (FISH), 0-1% by Immunohistochemistry (IHC), or 2+ by IHC and no evidence of amplification by FISH.

Exclusion Criteria:

* Treatment with another chemotherapy or hormonal therapy within the past 2 weeks.
* Treatment with trastuzumab, bevacizumab or other targeted therapies within the past 2 weeks.
* Concurrent treatment with radiotherapy.
* Ongoing treatment with any other investigational therapy.
* Prior treatment with eribulin
* Severe, concurrent illness including congestive heart failure, significant cardiac disease and uncontrolled hypertension, that would likely prevent the patient from being able to comply with the study protocol.
* Inadequate bone marrow, renal, or hepatic function as defined above, or an active coagulopathy that precludes tissue biopsy.
* Pregnant or lactating women and women of child-bearing potential who are not using an effective method of birth control. Women of childbearing potential must undergo a serum pregnancy test within seven days of starting the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-07-12 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2019-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope S. Rugo, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Duke University Cancer Center, Durham, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase Ib/1: 600 mg/Day PLX3397 Combined With Eribulin; Phase Ib/3: 600 mg/Day PLX3397 Combined With Eribulin: Treatments were given in 21 day Cycles. For each cycle, participants received 600 mg/day of PLX3397 in 100-200 mg gelcaps, by mouth daily & Eribulin 1.4 mg/m2 intravenously on days 1 and 8.
- Phase Ib/2: 400 mg/Day PLX3397 Combined With Eribulin: Treatments were given in 21 day Cycles. For each cycle, participants received 400 mg/day of PLX3397 in 100-200 mg gelcaps, by mouth daily & Eribulin 1.1 mg/m2 intravenously on days 1 and 8.
- Phase Ib/4: 800 mg/Day PLX3397 Combined With Eribulin; Phase Ib/5: 800 mg/Day PLX3397 Combined With Eribulin: Treatments were given in 21 day Cycles. For each cycle, participants received 800 mg/day of PLX3397 in 100-200 mg gelcaps, by mouth daily & Eribulin 1.4 mg/m2 intravenously on days 1 and 8.
- Phase Ib/6: 1000 mg/Day PLX3397 Combined With Eribulin: Treatments were given in 21 day Cycles. For each cycle, participants received 1000 mg/day of PLX3397 in 100-200 mg gelcaps, by mouth daily & Eribulin 1.4 mg/m2 intravenously on days 1 and 8.
- Phase II/1: 1000 mg/Day PLX3397 Combined With Eribulin: Treatment began with a 7 day Lead-in Phase, consisting of 1000 mg/day PLX3397 given by mouth for 5 days followed by 2 days of rest (no PLX3397). Then combination treatment was given in 21 day cycles. For each cycle, participants received 1000 mg/day of PLX3397 by mouth in the form of 100-200 mg gelcaps for 5 days followed by 2 days of rest repeated weekly and Eribulin at 1.4 mg/m2 intravenously on days 1 and 8.
- Phase II/2: 800 mg/Day PLX3397 Lead In+Combined With Eribulin: Treatment began with a 7 day Lead-in Phase, consisting of 800 mg/day PLX3397 given by mouth for 5 days followed by 2 days of rest (no PLX3397). Then combination treatment was given in 21 day cycles. For each cycle, participants received 800 mg/day of PLX3397 by mouth in the form of 100-200 mg gelcaps for 5 days followed by 2 days of rest repeated weekly and Eribulin at 1.4 mg/m2 intravenously on days 1 and 8.
Period: Overall Study
Arm/Group | Phase Ib/1: 600 mg/Day PLX3397 Combined With Eribulin | Phase Ib/2: 400 mg/Day PLX3397 Combined With Eribulin | Phase Ib/3: 600 mg/Day PLX3397 Combined With Eribulin | Phase Ib/4: 800 mg/Day PLX3397 Combined With Eribulin | Phase Ib/5: 800 mg/Day PLX3397 Combined With Eribulin | Phase Ib/6: 1000 mg/Day PLX3397 Combined With Eribulin | Phase II/1: 1000 mg/Day PLX3397 Combined With Eribulin | Phase II/2: 800 mg/Day PLX3397 Lead In+Combined With Eribulin
Started | 5 | 4 | 3 | 6 | 4 | 6 | 17 | 22
Completed | 5 | 4 | 3 | 6 | 4 | 6 | 17 | 22
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase II/2: 800 mg/Day PLX3397 Combined With Eribulin: Treatment began with a 7 day Lead-in Phase, consisting of 800 mg/day PLX3397 given by mouth for 5 days followed by 2 days of rest (no PLX3397). Then combination treatment was given in 21 day cycles. For each cycle, participants received 800 mg/day of PLX3397 by mouth in the form of 100-200 mg gelcaps for 5 days followed by 2 days of rest repeated weekly and Eribulin at 1.4 mg/m2 intravenously on days 1 and 8.
- Total: Total of all reporting groups
Arm/Group | Phase Ib/1: 600 mg/Day PLX3397 Combined With Eribulin | Phase Ib/2: 400 mg/Day PLX3397 Combined With Eribulin | Phase Ib/3: 600 mg/Day PLX3397 Combined With Eribulin | Phase Ib/4: 800 mg/Day PLX3397 Combined With Eribulin | Phase Ib/5: 800 mg/Day PLX3397 Combined With Eribulin | Phase Ib/6: 1000 mg/Day PLX3397 Combined With Eribulin | Phase II/1: 1000 mg/Day PLX3397 Combined With Eribulin | Phase II/2: 800 mg/Day PLX3397 Combined With Eribulin | Total
Number analyzed (Participants) | 5 | 4 | 3 | 6 | 4 | 6 | 17 | 22 | 67
Age, Continuous [Median (Full Range); unit: years] | 50.79 [33.2 to 60.5] | 54.38 [39.1 to 67.9] | 41.88 [39.5 to 46.4] | 51.30 [37.0 to 63.6] | 46.46 [36.7 to 60.0] | 48.33 [32.3 to 61.5] | 54.31 [39.7 to 71.1] | 56.06 [37.9 to 79.7] | 51.54 [32.3 to 79.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 3 | 6 | 4 | 6 | 17 | 22 | 67
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 7
  Not Hispanic or Latino | 4 | 3 | 3 | 3 | 4 | 6 | 14 | 18 | 55
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  White | 4 | 3 | 1 | 4 | 3 | 4 | 12 | 14 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 1 | 4 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of PLX3397 Given in Combination With Standard Dose Eribulin in Participants With Metastatic Breast Cancer (Phase 1b)
Description: The MTD was determined using a standard dose-escalation schema with 3 to 6 participants per cohort (3+3 design) for participants enrolled in Phase 1b. The starting dose level of PLX3397 was 600 mg/day and was raised in successive cohorts up to a dose of 1000 mg/day. Participants in each Phase Ib cohort were followed for dose limiting toxicities (DLTs) within the first 21 days of combination therapy and had to receive at least 14 days of PLX3397 and 2 doses of eribulin during the first cycle in order to be considered evaluable for DLT (unless the missed doses were due to a DLT). A toxicity was considered a DLT if it was treatment related and met specific requirements for type of toxicity and severity assessed according to Common Terminology Criteria for Adverse Events (CTCAE) version 4. The MTD was defined as the lowest dose level at which 2 or more participants in a cohort experienced a DLT. The dose level just below the MTD was selected for Phase 2.
Time Frame: Up to Day 21
Measure: Number; unit: miligrams per day
Groups:
- Phase Ib: Eribulin in Combination With PLX3397: Phase Ib:
  21 day treatment cycle: PLX3397 100-200 mg gelcaps, by mouth daily & Eribulin 1.4 mg/m2 intravenously, day 1 and 8
  * Cohort 1: 600 mg/day
  * Cohort 2: 800 mg/day
  * Cohort 3: 1000 mg/day
Arm/Group | Phase Ib: Eribulin in Combination With PLX3397
Number analyzed (Participants) | 28
miligrams per day | 1,000

2. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs) (Phase Ib)
Description: DLTs are select treatment related toxicities described in the protocol that were Grade 3 or 4 in severity per CTCAE v4, occurring within the first 21 days of combination therapy for patients enrolled in Phase Ib (for example, Grade 3 thrombocytopenia with significant bleeding, Grade 4 neutropenia lasting more than 5 days, or any Grade 3 or higher non-hematologic toxicity other than alopecia unless clearly unrelated to treatment). Grade 3 and 4 toxicities are considered severe and may be life threatening. Participants had to receive at least 14 days of PLX3397 and 2 doses of eribulin during the first cycle in order to be considered evaluable for DLT (unless the missed doses were due to a DLT). A treatment delay of greater than 7 days for PLX3397 or inability to get two doses of eribulin in the first cycle due to toxicity that was unrelated to cancer worsening or other illness was considered a DLT.
Time Frame: Up to Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib/1: 600 mg/Day PLX3397 Combined With Eribulin | Phase Ib/2: 400 mg/Day PLX3397 Combined With Eribulin | Phase Ib/3: 600 mg/Day PLX3397 Combined With Eribulin | Phase Ib/4: 800 mg/Day PLX3397 Combined With Eribulin | Phase Ib/5: 800 mg/Day PLX3397 Combined With Eribulin | Phase Ib/6: 1000 mg/Day PLX3397 Combined With Eribulin
Number analyzed (Participants) | 5 | 4 | 3 | 6 | 4 | 6
Participants | 3 | 0 | 0 | 1 | 0 | 1

3. Primary Outcome: Percentage of Total Phase II Participants With Chemotherapy Pre-Treated Triple Negative Metastatic Breast Cancer Who Are Progression Free at 3 Months
Description: Progression-free survival (PFS) at 3 months is defined as the proportion of participants in the combined Phase II cohorts that are alive and progression-free 90 days after Study Day 1, from the first administration of PLX3397 with eribulin. Duration of PFS is defined as the time from Study Day 1 to the earlier of disease progression or death due to any cause. These analyses are designed to include only objective progression events per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. PFS will be estimated as a simple percentage based upon the results of the 3 month tumor assessment. Participants for whom this assessment is not performed will be included as failures, even if known to be alive at this time point. Confidence intervals will be provided.
Time Frame: Up to 3 months
Population: Both Phase II Cohorts were combined for this planned analysis. Only 31 participants in Phase II obtained an objective progression event per RECIST v1.1 criteria at month 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Phase II: PLX3397 Combined With Eribulin: Treatment began with a 7 day Lead-in Phase, consisting of 800 mg or 1000 mg/day PLX3397 given by mouth for 5 days followed by 2 days of rest (no PLX3397). Then combination treatment was given in 21 day cycles. For each cycle, participants received 800 mg or 1000mg /day of PLX3397 by mouth in the form of 100-200 mg gelcaps for 5 days followed by 2 days of rest repeated weekly and Eribulin at 1.4 mg/m2 intravenously on days 1 and 8.
Arm/Group | Phase II: PLX3397 Combined With Eribulin
Number analyzed (Participants) | 31
Percentage of Participants | 35.7 [21.5 to 59.4]

4. Secondary Outcome: Objective Response Rate (ORR) (Phase II)
Description: The objective response rate (ORR) is defined as the proportion of patients for whom the best overall response at the time of data cutoff is confirmed complete response (CR) or confirmed partial response (PR) as assessed per Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 criteria. The analysis of ORR employed the Per Protocol population. Patients who did not have any post-baseline tumor assessments were counted as non-responders.
Time Frame: From baseline until study completion, an average of 24 months
Population: Both Phase II Cohorts were combined for this planned analysis. Only 31 participants in Phase II obtained an objective event per RECIST v1.1
Measure: Number; unit: percentage of participants
Arm/Group | Phase II: PLX3397 Combined With Eribulin
Number analyzed (Participants) | 31
percentage of participants | 16

5. Secondary Outcome: Median Duration of Response (Phase II)
Description: Duration of response is defined as the time from first documentation of objective response that is subsequently confirmed to progressive disease (PD) by the criteria or death due to any cause. Responders who have not been documented to have progressed or died at time of data cutoff will be right censored at the last available adequate tumor assessment. Median duration of response and its associated confidence interval will be estimated using the Kaplan-Meier method.
Time Frame: From date of first confirmed disease response to confirmed disease progression or death due to any cause, an average of 2 months
Population: Both Phase II Cohorts were combined for this planned analysis. Only 5 participants in Phase II obtained an objective response
Measure: Median (Full Range); unit: days
Arm/Group | Phase II: PLX3397 Combined With Eribulin
Number analyzed (Participants) | 5
days | 94 [46 to 130]

6. Secondary Outcome: Median Time to Disease Progression (Phase II)
Description: Time to progression will be estimated using the Kaplan-Meier method. Efficacy responses, disease progression and relapse classified based on RECIST v1.1 criteria will be used to determine progression. Time to progression will be calculated from the first administration of PLX3397 with eribulin. Participants who do not have disease progression will be censored at the date of the last evaluation for study disease or at the time of initiation of the new therapy, whichever is earlier. Patients lacking any response assessment after randomization will be censored at Day 1
Time Frame: From Day 1 to date of disease progression, an average of 4 months
Population: Both Phase II Cohorts were combined for this planned analysis. Only 31 participants in Phase II obtained an objective progression event per RECIST v1.1 criteria
Measure: Median (Full Range); unit: days
Arm/Group | Phase II: PLX3397 Combined With Eribulin
Number analyzed (Participants) | 31
days | 50.2 [21 to 230]

ADVERSE EVENTS:
Time Frame: Up to 24 months
Groups:
- Phase Ib/1: 600 mg/Day PLX3397 Combined With Eribulin: Treatments are given in 21 day cycles. For each cycle, treatment includes:
  * PLX3397 at a dose of 600 mg/day taken by mouth in the form of 100-200 mg gelcaps
  * Eribulin at dose of 1.4 mg/m2 given intravenously on days 1 and 8.
  PLX3397: Dosage Form: 100 mg or 200 mg capsules, Dosage: 600mg, oral administration
  Eribulin: Dosage Form: 1 mg per 2 mL (0.5 mg per mL); Solution (clear, colorless, sterile, packaged in glass vial) Dosage: 1.4 mg/m2, 2-5 min IV, Day 1, 8 q21 days
- Phase Ib/2: 400 mg/Day PLX3397 Combined With Eribulin: Treatments are given in 21 day cycles. For each cycle, treatment includes:
  * PLX3397 at a dose of 400 mg/day taken by mouth in the form of 100-200 mg gelcaps
  * Eribulin at dose of 1.4 mg/m2 given intravenously on days 1 and 8.
  PLX3397: Dosage Form: 100 mg or 200 mg capsules, Dosage: 400mg, oral administration
  Eribulin: Dosage Form: 1 mg per 2 mL (0.5 mg per mL); Solution (clear, colorless, sterile, packaged in glass vial) Dosage: 1.4 mg/m2, 2-5 min IV, Day 1, 8 q21 days
- Phase Ib/3: 600 mg/Day PLX3397 Combined With Eribulin: Treatments are given in 21 day cycles. For each cycle, treatment includes:
  * PLX3397 at a dose of 600 mg/day taken by mouth in the form of 100-200 mg gelcaps
  * Eribulin at dose of 1.4 mg/m2 given intravenously on days 1 and 8.
  PLX3397: Dosage Form: 100 mg or 200 mg capsules, Dosage: 600 mg, oral administration
  Eribulin: Dosage Form: 1 mg per 2 mL (0.5 mg per mL); Solution (clear, colorless, sterile, packaged in glass vial) Dosage: 1.4 mg/m2, 2-5 min IV, Day 1, 8 q21 days
- Phase Ib/4: 800 mg/Day PLX3397 Combined With Eribulin; Phase Ib/5: 800 mg/Day PLX3397 Combined With Eribulin: Treatments are given in 21 day cycles. For each cycle, treatment includes:
  * PLX3397 at a dose of 800 mg/day taken by mouth in the form of 100-200 mg gelcaps
  * Eribulin at dose of 1.4 mg/m2 given intravenously on days 1 and 8
  PLX3397: Dosage Form: 100 mg or 200 mg capsules, Dosage: 800 mg, oral administration
  Eribulin: Dosage Form: 1 mg per 2 mL (0.5 mg per mL); Solution (clear, colorless, sterile, packaged in glass vial) Dosage: 1.4 mg/m2, 2-5 min IV, Day 1, 8 q21 days
- Phase Ib/6: 1000 mg/Day PLX3397 Combined With Eribulin: Treatments are given in 21 day cycles. For each cycle, treatment includes:
  * PLX3397 at a dose of 1000 mg/day taken by mouth in the form of 100-200 mg gelcaps
  * Eribulin at dose of 1.4 mg/m2 given intravenously on days 1 and 8
  PLX3397: Dosage Form: 100 mg or 200 mg capsules, Dosage: 1000 mg, oral administration
  Eribulin: Dosage Form: 1 mg per 2 mL (0.5 mg per mL); Solution (clear, colorless, sterile, packaged in glass vial) Dosage: 1.4 mg/m2, 2-5 min IV, Day 1, 8 q21 days
- Phase II/1: 1000 mg/Day PLX3397 Combined With Eribulin: Treatment begins with a 7 day Lead-in phase of PLX3397 alone, followed by 21 day cycles of PLX3397 in combination with eribulin.
  Lead-in phase treatment:
  * PLX3397 at a dose of 1000 mg/day given by mouth in the form of 100-200 mg gelcaps for 5 days followed by 2 days of rest.
  Treatment given in each 21 day cycle:
  * PLX3397 at a dose of 1000 mg/day given by mouth in the form of 100-200 mg gelcaps for 5 days followed by 2 days of rest, repeated weekly
  * Eribulin at dose of 1.4 mg/m2 given intravenously on days 1 and 8
  PLX3397: Dosage Form: 100 mg or 200 mg capsules, Dosage: 1000 mg, oral administration
  Eribulin: Dosage Form: 1 mg per 2 mL (0.5 mg per mL); Solution (clear, colorless, sterile, packaged in glass vial) Dosage: 1.4 mg/m2, 2-5 min IV, Day 1, 8 q21 days
- Phase II/2: 800 mg/Day PLX3397 Combined With Eribulin: Treatment begins with a 7 day Lead-in phase of PLX3397 alone, followed by 21 day cycles of PLX3397 in combination with eribulin.
  Lead-in phase treatment:
  * PLX3397 at a dose of 800 mg/day given by mouth in the form of 100-200 mg gelcaps for 5 days followed by 2 days of rest.
  Treatment given in each 21 day cycle:
  * PLX3397 at a dose of 800 mg/day given by mouth in the form of 100-200 mg gelcaps for 5 days followed by 2 days of rest, repeated weekly
  * Eribulin at dose of 1.4 mg/m2 given intravenously on days 1 and 8
  PLX3397: Dosage Form: 100 mg or 200 mg capsules, Dosage: 800 mg, oral administration
  Eribulin: Dosage Form: 1 mg per 2 mL (0.5 mg per mL); Solution (clear, colorless, sterile, packaged in glass vial) Dosage: 1.4 mg/m2, 2-5 min IV, Day 1, 8 q21 days
Arm/Group | Phase Ib/1: 600 mg/Day PLX3397 Combined With Eribulin | Phase Ib/2: 400 mg/Day PLX3397 Combined With Eribulin | Phase Ib/3: 600 mg/Day PLX3397 Combined With Eribulin | Phase Ib/4: 800 mg/Day PLX3397 Combined With Eribulin | Phase Ib/5: 800 mg/Day PLX3397 Combined With Eribulin | Phase Ib/6: 1000 mg/Day PLX3397 Combined With Eribulin | Phase II/1: 1000 mg/Day PLX3397 Combined With Eribulin | Phase II/2: 800 mg/Day PLX3397 Combined With Eribulin
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/3 | 1/6 | 0/4 | 0/6 | 1/17 | 0/22
Serious Adverse Events (participants affected / at risk) | 3/5 | 3/4 | 1/3 | 2/6 | 1/4 | 3/6 | 6/17 | 14/22
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 1/3 | 4/6 | 3/4 | 6/6 | 14/17 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib/1: 600 mg/Day PLX3397 Combined With Eribulin (N=5) | Phase Ib/2: 400 mg/Day PLX3397 Combined With Eribulin (N=4) | Phase Ib/3: 600 mg/Day PLX3397 Combined With Eribulin (N=3) | Phase Ib/4: 800 mg/Day PLX3397 Combined With Eribulin (N=6) | Phase Ib/5: 800 mg/Day PLX3397 Combined With Eribulin (N=4) | Phase Ib/6: 1000 mg/Day PLX3397 Combined With Eribulin (N=6) | Phase II/1: 1000 mg/Day PLX3397 Combined With Eribulin (N=17) | Phase II/2: 800 mg/Day PLX3397 Combined With Eribulin (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft Tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and Infestations other (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient Ischemia Attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib/1: 600 mg/Day PLX3397 Combined With Eribulin (N=5) | Phase Ib/2: 400 mg/Day PLX3397 Combined With Eribulin (N=4) | Phase Ib/3: 600 mg/Day PLX3397 Combined With Eribulin (N=3) | Phase Ib/4: 800 mg/Day PLX3397 Combined With Eribulin (N=6) | Phase Ib/5: 800 mg/Day PLX3397 Combined With Eribulin (N=4) | Phase Ib/6: 1000 mg/Day PLX3397 Combined With Eribulin (N=6) | Phase II/1: 1000 mg/Day PLX3397 Combined With Eribulin (N=17) | Phase II/2: 800 mg/Day PLX3397 Combined With Eribulin (N=22)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 3 (6) | 2 (2) | 7 (18) | 8 (24)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (7) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 2 (3) | 3 (7) | 2 (3) | 7 (20) | 10 (24)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (5) | 1 (2) | 1 (1) | 0 (0) | 2 (5) | 1 (1) | 9 (23) | 7 (18)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
White blood cell decreased (Investigations) | 3 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (12) | 2 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (5) | 7 (7)
Mucositis oral (Gastrointestinal disorders) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 9 (11) | 8 (11)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (13)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Fatigue (General disorders) | 3 (4) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 10 (13) | 14 (19)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 6 (7) | 5 (21)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 0 (0) | 3 (4) | 1 (3) | 1 (3) | 5 (12) | 7 (15)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (5) | 4 (5) | 3 (3)
Hpyerglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (9)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 6 (7) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 3 (7)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 6 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 5 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (6)
Anzxiety (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Hepatic Failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT01596751/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT01596751/ICF_001.pdf